CLINICAL TRIAL: NCT01353508
Title: A Randomized, Double-blind, Controlled, Crossover Study to Evaluate the Sodium Excretion of LCZ696 in Patients With Stable Heart Failure, in Patients With Hypertension, and in Healthy Volunteers
Brief Title: Sodium Excretion of LCZ696 in Patients With Hypertension; Heart Failure and Healthy Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLCZ696B2223
Record Dates: First submitted 2011-03-16; First posted 2011-05-13 (Estimated); Results first posted 2015-11-23 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-10

CONDITIONS: Hypertension
Keywords: Sodium excretion,; LCZ696
MeSH Terms: conditions — Hypertension | interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- LCZ696 to Valsartan - Heart Failure (HF) cohort (Experimental): Participants in this arm received Valsartan 160 mg twice daily (bid) during open-label run-in, LCZ696 200 mg bid double blind treatment during period 1, Valsartan 160 mg bid during wash-out, and Valsartan 160 mg bid double blind treatment during period 2.
  Interventions: Drug: LCZ696; Drug: Valsartan
- Valsartan to LCZ696 - HF Cohort (Experimental): Participants in this arm received Valsartan 160 mg twice daily bid during open-label run-in, Valsartan 160 mg bid during period 1, Valsartan 160 mg bid during wash-out, and LCZ696 200 mg bid double blind treatment during period 2.
  Interventions: Drug: LCZ696; Drug: Valsartan
- LCZ696 to Valsartan - Hypertension (HTN) cohort (Experimental): Participants in this arm received Valsartan 320 mg once daily (qd) during open-label run-in, LCZ696 400 mg qd double blind treatment during period 1, Valsartan 320 mg qd during wash-out, and Valsartan 320 mg qd double blind treatment during period 2.
  Interventions: Drug: LCZ696; Drug: Valsartan
- Valsartan to LCZ696 - HTN cohort (Experimental): Participants in this arm received Valsartan 320 mg qd during open-label run-in, Valsartan 320 mg qd during period 1, Valsartan 320 mg qd during wash-out, and LCZ696 400 qd bid double blind treatment during period 2.
  Interventions: Drug: LCZ696; Drug: Valsartan

INTERVENTIONS:
Drug: LCZ696 — 200 mg and 400 mg tablets
Drug: Valsartan — 160 mg tablets

SUMMARY:
Assess mechanism of action of LCZ696 related to sodium excretion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart failure: documented NYHA class II-III heart failure
* Patients with hypertension: stable hypertensive medication for the preceding 2 months

Exclusion Criteria:

* Women of childbearing potential
* History of recent myocardial infarction
* History of dialysis or renal transplant
* Patients with type 1 diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Moscow, Russia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In each of the HF and HTN cohorts, 16 participants (total = 32) received LCZ696 or Valsartan in period 1. Then, there was a cross-over where participants received LCZ96 or Valsartan in period 2.
Period: Period 1 - First Intervention (7 Days)
Arm/Group | LCZ696 to Valsartan - Heart Failure (HF) Cohort | Valsartan to LCZ696 - HF Cohort | LCZ696 to Valsartan - Hypertension (HTN) Cohort | Valsartan to LCZ696 - HTN Cohort
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 7
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Period 2 - Second Intervention (7 Days)
Arm/Group | LCZ696 to Valsartan - Heart Failure (HF) Cohort | Valsartan to LCZ696 - HF Cohort | LCZ696 to Valsartan - Hypertension (HTN) Cohort | Valsartan to LCZ696 - HTN Cohort
Started | 8 | 8 | 8 | 7
Completed | 7 | 8 | 8 | 7
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCZ696 to Valsartan - Heart Failure (HF) Cohort | Valsartan to LCZ696 - HF Cohort | LCZ696 to Valsartan - Hypertension (HTN) Cohort | Valsartan to LCZ696 - HTN Cohort | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age mean and standard deviation (SD) for HF cohort was 65.4 (9.57); age mean and SD for HTN cohort was 58.8 (8.15)
  Years | 63.3 (10.15) | 67.6 (9.07) | 58.0 (8.02) | 61.6 (8.40) | 62.6 (8.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 5 | 2 | 9
  Male | 6 | 8 | 3 | 6 | 23

OUTCOME MEASURES:

1. Primary Outcome: 24-hour Urinary Sodium Excretion
Description: Urine was collected in 12-hour intervals, and of each pooled 24-hour (daily) sample, sodium concentration was measured. The measure type used for this outcome measure (OM) was Geometric Least square Means (LSM).
Time Frame: day 1
Population: The Pharmacodynamic (PD) analysis set, which included all participants who had no major protocol deviation with impact on PD data, were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/24 hours
Groups:
- LCZ696 - Heart Failure (HF) Cohort: Participants in this arm received Valsartan 160 mg twice daily (bid) during open-label run-in, LCZ696 200 mg bid double blind treatment during period 1, Valsartan 160 mg bid during wash-out, and Valsartan 160 mg bid double blind treatment during period 2.
- Valsartan - HF Cohort: Participants in this arm received Valsartan 160 mg twice daily bid during open-label run-in, Valsartan 160 mg bid during period 1, Valsartan 160 mg bid during wash-out, and LCZ696 200 mg bid double blind treatment during period 2.
- LCZ696 - Hypertension (HTN) Cohort: Participants in this arm received Valsartan 320 mg once daily (qd) during open-label run-in, LCZ696 400 mg qd double blind treatment during period 1, Valsartan 320 mg qd during wash-out, and Valsartan 320 mg qd double blind treatment during period 2.
- Valsartan - HTN Cohort: Participants in this arm received Valsartan 320 mg qd during open-label run-in, Valsartan 320 mg qd during period 1, Valsartan 320 mg qd during wash-out, and LCZ696 400 qd bid double blind treatment during period 2.
Arm/Group | LCZ696 - Heart Failure (HF) Cohort | Valsartan - HF Cohort | LCZ696 - Hypertension (HTN) Cohort | Valsartan - HTN Cohort
Number analyzed (Participants) | 16 | 16 | 16 | 16
mmol/24 hours | 220.58 [182.64 to 266.41] | 198.73 [163.50 to 241.56] | 177.40 [152.65 to 206.15] | 146.18 [126.42 to 169.03]

2. Primary Outcome: Cumulative 7-day Urinary Sodium Excretion
Description: as for outcome 1
Time Frame: 7 day-cummulative (days 1 through 7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/7 days
Arm/Group | LCZ696 - Heart Failure (HF) Cohort | Valsartan - HF Cohort | LCZ696 - Hypertension (HTN) Cohort | Valsartan - HTN Cohort
Number analyzed (Participants) | 16 | 16 | 16 | 16
mmol/7 days | 1020.57 [903.47 to 1152.84] | 1114.18 [983.37 to 1262.39] | 906.81 [839.94 to 979.00] | 943.26 [873.62 to 1018.45]

3. Secondary Outcome: 24-hour Diuresis
Description: Urine was collected in 12-hour intervals, and of each pooled 24-hour (daily) sample, urine volume was measured. The measure type used for this OM was Geometric LSM.
Time Frame: day 1
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/24 hours
Arm/Group | LCZ696 - Heart Failure (HF) Cohort | Valsartan - HF Cohort | LCZ696 - Hypertension (HTN) Cohort | Valsartan - HTN Cohort
Number analyzed (Participants) | 16 | 16 | 16 | 16
mL/24 hours | 3199.37 [2662.17 to 3844.96] | 2874.36 [2375.61 to 3477.82] | 3382.94 [2859.86 to 4001.70] | 2393.61 [2034.84 to 2815.64]

4. Secondary Outcome: 7-day Cumulative Diuresis
Description: as for outcome 3
Time Frame: 7-day cumulative (days 1 through 7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | LCZ696 - Heart Failure (HF) Cohort | Valsartan - HF Cohort | LCZ696 - Hypertension (HTN) Cohort | Valsartan - HTN Cohort
Number analyzed (Participants) | 16 | 16 | 16 | 16
mL | 12347.92 [10842.81 to 14062.48] | 13180.02 [11539.55 to 15053.71] | 16980.05 [15627.59 to 18449.54] | 15265.35 [14048.28 to 16587.87]

5. Secondary Outcome: Urinary Cyclic Guanosine Monophosphate (cGMP) Excretion Over 24 Hours
Description: cGMP was analyzed at a central laboratory. The measure type used for this OM was Geometric LSM.
Time Frame: day 1, day 6, day 7
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: nmol/24 hours
Arm/Group | LCZ696 - Heart Failure (HF) Cohort | Valsartan - HF Cohort | LCZ696 - Hypertension (HTN) Cohort | Valsartan - HTN Cohort
Number analyzed (Participants) | 16 | 16 | 16 | 16
nmol/24 hours
  Day 1 | 1851.79 [1504.96 to 2278.56] | 884.99 [713.93 to 1097.03] | 1085.76 [867.64 to 1358.71] | 557.53 [448.87 to 692.51]
  Day 6 | 1467.67 [1153.25 to 1867.79] | 865.62 [674.39 to 1111.07] | 863.32 [707.64 to 1053.25] | 562.11 [460.85 to 685.63]
  Day 7 | 1571.02 [1331.84 to 1853.15] | 859.07 [723.03 to 1020.72] | 1107.04 [869.95 to 1408.76] | 603.90 [474.68 to 768.30]

6. Secondary Outcome: Percent Change From Baseline in Plasma Mid-regional Pro-atrial Natriuretic Peptide (MR-proANP) Biomarker
Description: MR-proANP was analyzed at a central laboratory.
Time Frame: 2, 4, 6 and 12 hours post dose on day 1; 24 hours post dose on day 2; 2, 4, 6 and 12 hours post dose on day 7
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | LCZ696 - Heart Failure (HF) Cohort | Valsartan - HF Cohort | LCZ696 - Hypertension (HTN) Cohort | Valsartan - HTN Cohort
Number analyzed (Participants) | 16 | 16 | 16 | 16
Percentage change
  Day 1, 2.0 hours post dose | -7.04 [-12.21 to -1.87] | 2.08 [-3.48 to 7.63] | -10.11 [-17.41 to -2.82] | -1.66 [-7.99 to 4.68]
  Day 1, 4.0 hrs post dose | -17.39 [-24.68 to -10.10] | -6.74 [-14.32 to 0.84] | -12.68 [-25.45 to 0.08] | -7.33 [-19.27 to 4.61]
  Day 1, 6.0 hours post dose | -23.99 [-31.64 to -16.33] | -10.16 [-18.08 to -2.23] | -17.82 [-25.16 to -10.48] | -4.52 [-11.60 to 2.56]
  Day 1, 12.0 hrs post dose | -27.58 [-38.93 to -16.22] | -7.48 [-19.26 to 4.29] | -19.77 [-32.56 to -6.98] | -15.20 [-27.10 to -3.31]
  Day 2, 24.0 hrs post dose | -25.13 [-35.53 to -14.73] | -14.53 [-25.28 to -3.78] | -17.30 [-33.46 to -1.13] | -9.45 [-24.39 to 5.50]
  Day 7, 0.0 hours | -21.27 [-29.72 to -12.81] | -2.54 [-11.30 to 6.21] | -16.03 [-28.52 to -3.53] | 0.44 [-11.59 to 12.46]
  Day 7, 4.0 hours post dose | -24.35 [-35.18 to -13.52] | 1.64 [-9.62 to 12.91] | -19.34 [-31.20 to -7.49] | -2.56 [-13.90 to 8.78]
  Day 7, 6.0 hours post dose | -23.40 [-33.98 to -12.82] | -3.53 [-14.54 to 7.48] | -20.84 [-33.62 to -8.05] | -1.98 [-14.25 to 10.28]
  Day 7, 12.0 hours post dose | -20.95 [-33.10 to -8.80] | -12.65 [-25.27 to -0.03] | -23.09 [-35.90 to -10.28] | -10.27 [-22.61 to 2.06]

7. Secondary Outcome: Percent Change From Baseline in Brain Natriuretic Peptide (BNP) Biomarker
Description: BNP was analyzed at a central laboratory.
Time Frame: 0.5, 1, 2, 4, 6 and 12 hours post dose on day 1; 24 hours post dose on day 2; 0, 4, 6 and 12 hours post dose on day 7
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | LCZ696 - Heart Failure (HF) Cohort | Valsartan - HF Cohort | LCZ696 - Hypertension (HTN) Cohort | Valsartan - HTN Cohort
Number analyzed (Participants) | 16 | 16 | 16 | 16
Percentage change
  Day 1, 0.5 hour post dose | 72.32 [-70.26 to 214.90] | -8.93 [-151.85 to 133.99] | -10.75 [-28.59 to 7.08] | -5.94 [-23.59 to 11.71]
  Day 1, 1.0 hr post dose | 121.85 [-86.02 to 329.72] | -0.83 [-209.19 to 207.53] | 1218.56 [-760.23 to 3197.35] | -33.19 [-1865.92 to 1799.53]
  Day 1, 2.0 hours post dose | 176.35 [-85.34 to 438.04] | 21.92 [-215.63 to 259.47] | 31.10 [8.44 to 53.76] | -0.38 [-21.37 to 20.61]
  Day 1, 4.0 hrs post dose | 50.12 [30.22 to 70.02] | -1.78 [-21.01 to 17.44] | 38.82 [18.71 to 58.92] | 11.06 [-7.56 to 29.68]
  Day 1, 6.0 hrs post dose | 130.62 [-10.46 to 271.70] | 11.09 [-130.33 to 152.51] | 68.23 [11.48 to 124.97] | 7.97 [-44.59 to 60.52]
  Day 1, 12.0 hrs post dose | 90.58 [28.51 to 152.66] | 30.07 [-32.15 to 92.29] | 85.93 [23.34 to 148.52] | 8.51 [-48.97 to 65.99]
  Day 2, 24 hrs post dose | 102.88 [-84.18 to 289.93] | 5.18 [-174.46 to 184.81] | -0.66 [-31.34 to 30.02] | -20.61 [-47.16 to 5.94]
  Day 7, 0.0 hr | 190.96 [-100.59 to 482.51] | 27.75 [-264.49 to 320.00] | 14.20 [-28.81 to 57.21] | -7.19 [-48.17 to 33.79]
  Day 7, 4.0 hrs post dose | 220.38 [-72.28 to 513.04] | 34.44 [-249.44 to 318.31] | 34.92 [-6.58 to 76.42] | 5.20 [-34.59 to 44.99]
  Day 7, 6.0 hrs post dose | 195.06 [-94.90 to 485.02] | 46.75 [-257.14 to 350.63] | 7.78 [-33.49 to 49.04] | 7.82 [-29.68 to 45.32]
  Day 7, 12.0 hrs post dose | 236.05 [-173.38 to 645.47] | 70.31 [-334.37 to 474.99] | 38.45 [-13.98 to 90.88] | 25.79 [-24.48 to 76.06]

8. Secondary Outcome: Percent Change From Baseline in Mid-regional Pro-adrenomedullin (MR-proADM) Biomarker
Description: MR-proADM was analyzed at a central laboratory.
Time Frame: 2, 4, 6 and 12 hours post dose on day 1; 24 hours post dose on day 2; 0, 4, 6 and 12 hours post dose on day 7
Population: The HF arms only of the Pharmacodynamic (PD) analysis set, which included all participants who had no major protocol deviation with impact on PD data, were included in the analysis. MR-proADM is considered a biomarker for HF only; therefore, the HTN cohort was not assessed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | LCZ696 - Heart Failure (HF) Cohort | Valsartan - HF Cohort
Number analyzed (Participants) | 16 | 16
Percentage change
  Day 1, 2.0 hours post dose | 8.04 [-0.34 to 16.42] | -2.87 [-11.53 to 5.79]
  Day 1, 4.0 hrs post dose | 21.22 [11.38 to 31.06] | -8.22 [-18.03 to 1.59]
  Day 1, 6.0 hrs post dose | 20.18 [10.05 to 30.31] | -8.81 [-18.90 to 1.27]
  Day 1, 12.0 hrs post dose | 40.70 [22.25 to 59.15] | 7.61 [-10.84 to 26.05]
  Day 2, 24 hrs post dose | 57.28 [42.29 to 72.26] | 0.72 [-14.26 to 15.70]
  Day 7, 0.0 hrs | 61.28 [47.35 to 75.21] | 1.38 [-12.07 to 14.83]
  Day 7, 4.0 hrs post dose | 51.71 [39.67 to 63.74] | -5.27 [-16.90 to 6.36]
  Day 7, 6.0 hrs post dose | 48.22 [36.26 to 60.19] | -3.63 [-14.89 to 7.64]
  Day 7, 12.0 hrs post dose | 69.45 [50.70 to 88.20] | 2.15 [-16.60 to 20.90]

9. Secondary Outcome: Percent Change From Baseline in C-type Natriuretic Peptide (proCNP) Biomarker
Description: ProCNP was analyzed at a central laboratory.
Time Frame: 2, 4, 6, 8 and 12 hours post dose on day 1; day 2; 0, 4, 6, 8 and 12 hours post dose on day 7
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | LCZ696 - Heart Failure (HF) Cohort | Valsartan - HF Cohort
Number analyzed (Participants) | 16 | 16
Percentage change
  Day 1, 2.0 hrs post dose | 0.35 [-6.33 to 7.03] | -1.01 [-8.16 to 6.13]
  Day 1, 4.0 hours post dose | 34.58 [19.36 to 49.79] | -6.02 [-22.28 to 10.25]
  Day 1, 6.0 hrs post dose | 67.85 [42.32 to 93.37] | -16.19 [-43.85 to 11.48]
  Day 1, 8.0 hrs post dose | 123.75 [87.53 to 159.98] | -9.87 [-48.59 to 28.86]
  Day 1, 12.0 hrs post dose | 190.36 [148.95 to 231.78] | 15.55 [-29.00 to 60.09]
  Day 2, 24 hrs post dose | 218.81 [163.62 to 274.01] | 4.99 [-54.79 to 64.78]
  Day 7, 0.0 hour | 244.20 [186.26 to 302.14] | 0.09 [-61.85 to 62.04]
  Day 7, 4.0 hours post dose | 216.61 [159.66 to 273.56] | -8.94 [-69.82 to 51.95]
  Day 7, 6.0 hrs post dose | 211.21 [151.36 to 271.07] | -18.17 [-82.15 to 45.82]
  Day 7, 8.0 hrs post dose | 241.99 [181.22 to 302.76] | -11.30 [-76.27 to 53.67]
  Day 7, 12.0 hrs post dose | 278.58 [214.45 to 342.71] | 0.88 [-67.68 to 69.44]

10. Secondary Outcome: Percent Change From Baseline in C-terminal-proendothelin-1 (CT-proET-1) Biomarker
Description: CT-proET-1 was analyzed at a central laboratory.
Time Frame: 12 hours post dose on day 1; 24 hours post dose on day 2; 0 and 12 hours post dose on day 7
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | LCZ696 - Heart Failure (HF) Cohort | Valsartan - HF Cohort | LCZ696 - Hypertension (HTN) Cohort | Valsartan - HTN Cohort
Number analyzed (Participants) | 16 | 16 | 16 | 16
Percentage change
  Day 1, 12.0 hours post dose | 36.39 [26.14 to 46.65] | 2.51 [-8.14 to 13.16] | 108.87 [5.82 to 211.92] | 54.07 [-38.42 to 146.57]
  Day 2, 24.0 hours post dose | 32.44 [19.41 to 45.47] | 11.41 [-2.76 to 25.59] | 123.45 [36.65 to 210.25] | 38.70 [-41.78 to 119.19]
  Day 7, 0.0 hour | 31.98 [19.53 to 44.42] | 0.62 [-11.85 to 13.09] | 94.76 [17.45 to 172.06] | 41.77 [-32.97 to 116.50]
  Day 7, 12.0 hours post dose | 41.75 [26.81 to 56.69] | 7.05 [-8.97 to 23.08] | 117.84 [30.76 to 204.92] | 61.90 [-22.40 to 146.20]

11. Secondary Outcome: Percent Change From Baseline in N-terminal-proBNP (NT-proBNP) Biomarker
Description: NT-proBNP was analyzed at a central laboratory.
Time Frame: 2, 4, 6 and 12 hours post dose on day 1; 24 hours post dose on day 2; 0, 4, 6 and 12 hours post dose on day 7
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | LCZ696 - Heart Failure (HF) Cohort | Valsartan - HF Cohort | LCZ696 - Hypertension (HTN) Cohort | Valsartan - HTN Cohort
Number analyzed (Participants) | 16 | 16 | 16 | 16
Percentage change
  Day 1, 2.0 hours post dose | 3.06 [-1.80 to 7.92] | 6.87 [1.87 to 11.88] | 5.10 [-1.10 to 11.31] | 8.32 [2.32 to 14.32]
  Day 1, 4.0 hours post dose | 2.68 [-5.30 to 10.66] | 13.21 [5.02 to 21.40] | 44.79 [-11.93 to 101.51] | 22.14 [-32.65 to 76.93]
  Day 1, 6.0 hours post dose | 3.71 [-8.15 to 15.57] | 21.70 [9.59 to 33.80] | 12.58 [-4.17 to 29.33] | 21.21 [5.03 to 37.39]
  Day 1, 12.0 hours post dose | 17.15 [-3.58 to 37.89] | 42.32 [20.94 to 63.70] | 61.46 [3.83 to 119.09] | 33.17 [-22.28 to 88.62]
  Day 2, 24 hours post dose | -21.85 [-35.37 to -8.33] | 23.51 [9.48 to 37.54] | 8.61 [-20.73 to 37.95] | -4.41 [-32.64 to 23.81]
  Day 7, 0.0 hour | -19.57 [-34.08 to -5.05] | 2.29 [-12.74 to 17.32] | -10.14 [-35.77 to 15.48] | -0.13 [-25.77 to 25.51]
  Day 7, 4.0 hours post dose | -14.60 [-30.67 to 1.47] | 14.85 [-1.78 to 31.49] | -8.10 [-35.21 to 19.01] | 19.83 [-7.29 to 46.95]
  Day 7, 6.0 hours post dose | -15.05 [-32.53 to 2.43] | 17.34 [-0.75 to 35.44] | -9.42 [-37.40 to 18.57] | 20.47 [-6.63 to 47.58]
  Day 7, 12.0 hours post dose | 1.37 [-22.83 to 25.56] | 46.05 [20.87 to 71.22] | 12.22 [-26.18 to 50.62] | 47.27 [8.85 to 85.68]

12. Secondary Outcome: Percent Change From Baseline in Aldosterone Biomarker
Description: Aldosterone was analyzed at a central laboratory.
Time Frame: 6 and 12 hours post dose on day 1; 24 hours post dose on day 2; 0, 6 and 12 hours post dose on day 7
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | LCZ696 - Heart Failure (HF) Cohort | Valsartan - HF Cohort | LCZ696 - Hypertension (HTN) Cohort | Valsartan - HTN Cohort
Number analyzed (Participants) | 16 | 16 | 16 | 16
Percentage change
  Day 1, 6.0 hours post dose | 71.15 [29.66 to 112.64] | -14.63 [-56.02 to 26.77] | 90.51 [-39.10 to 220.12] | 72.92 [-48.38 to 194.22]
  Day 1, 12.0 hours post dose | 208.06 [44.03 to 372.10] | 8.36 [-155.05 to 171.77] | 249.13 [4.30 to 493.96] | 325.31 [96.75 to 553.86]
  Day 2, 24.0 hours post dose | 168.32 [65.01 to 271.63] | 71.73 [-35.08 to 178.55] | 438.28 [-67.61 to 944.17] | 524.93 [55.45 to 994.41]
  Day 7, 0.0 hour | 111.21 [16.31 to 206.11] | 21.68 [-77.33 to 120.69] | 49.91 [-12.58 to 112.40] | 5.61 [-55.0 to 66.22]
  Day 7, 6.0 hours post dose | 65.22 [7.48 to 122.95] | 24.58 [-31.70 to 80.87] | 24.47 [-104.07 to 153.01] | 107.60 [-16.47 to 231.67]
  Day 7, 12.0 hours post dose | 238.32 [-46.10 to 522.74] | 230.06 [-58.04 to 518.17] | 147.89 [-4.40 to 300.19] | 152.37 [4.74 to 300.00]

13. Secondary Outcome: Percent Change From Baseline in Urinary Electrolyte Excretion (Sodium, Potassium, Chloride and Calcium)
Description: Urine was collected in 12-hour intervals, and of each pooled 24-hour (daily) sample, sodium, potassium, albumin and calcium were measured.
Time Frame: 2, 4, 6 and 12 hours post dose on day 1; 24 hours post dose on day 2; 0, 4, 6 and 12 hours post dose on day 7
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | LCZ696 - Heart Failure (HF) Cohort | Valsartan - HF Cohort | LCZ696 - Hypertension (HTN) Cohort | Valsartan - HTN Cohort
Number analyzed (Participants) | 16 | 16 | 16 | 16
Percentage change
  Calcium, day 1, 2.0 hours post dose | -0.05 [-1.24 to 1.13] | -1.40 [-2.62 to -0.17] | 0.51 [-1.00 to 2.01] | 0.08 [-1.38 to 1.53]
  Calcium, day 1, 4.0 hours post dose | -2.19 [-3.78 to -0.60] | -2.46 [-4.11 to -0.81] | 0.76 [-1.39 to 2.91] | 0.27 [-1.79 to 2.33]
  Calcium, day 1, 6.0 hours post dose | -3.69 [-5.19 to -2.19] | -4.03 [-5.59 to -2.48] | -2.22 [-3.89 to -0.55] | -2.49 [-4.10 to -0.89]
  Calcium, day 1, 12.0 hours post dose | -2.80 [-4.24 to -1.37] | -1.34 [-2.83 to 0.16] | 1.77 [-0.40 to 3.94] | 0.82 [-1.27 to 2.91]
  Calcium, day 2, 24 hours post dose | -2.09 [-4.21 to 0.02] | 0.44 [-1.72 to 2.60] | 2.06 [-0.42 to 4.55] | 1.34 [-1.06 to 3.73]
  Calcium, day 7, 0.0 hour | -0.34 [-2.75 to 2.07] | -1.11 [-3.60 to 1.38] | -5.82 [-8.28 to -3.36] | -6.19 [-8.65 to -3.73]
  Calcium, day 7, 4.0 hours post dose | -2.45 [-4.09 to -0.81] | -2.17 [-3.87 to -0.47] | -8.46 [-10.95 to -5.98] | -7.42 [-9.90 to -4.94]
  Calcium, day 7, 6.0 hours post dose | -4.30 [-5.65 to -2.95] | -3.53 [-4.93 to -2.12] | -9.12 [-11.54 to -6.70] | -9.89 [-12.32 to -7.47]
  Calcium, day 7, 12.0 hours post dose | -3.41 [-4.94 to -1.88] | -1.27 [-2.86 to 0.32] | -4.63 [-6.89 to -2.36] | -4.99 [-7.25 to -2.73]
  Chloride, day 1, 2.0 hours post dose | -0.33 [-1.05 to 0.39] | -0.47 [-1.22 to 0.28] | -0.35 [-0.96 to 0.27] | 0.22 [-0.38 to 0.81]
  Chloride, day 1, 4.0 hours post dose | -1.35 [-2.07 to -0.64] | -0.61 [-1.36 to 0.14] | 0.05 [-0.62 to 0.72] | 0.41 [-0.23 to 1.05]
  Chloride, day 1, 6.0 hours post dose | -0.66 [-1.35 to 0.03] | -0.42 [-1.14 to 0.30] | -0.48 [-1.15 to 0.19] | 0.05 [-0.59 to 0.70]
  Chloride, day 1, 12.0 hours post dose | 0.46 [-0.49 to 1.41] | 1.44 [0.45 to 2.42] | -0.93 [-1.70 to -0.16] | -0.15 [-0.92 to 0.62]
  Chloride, day 2, 24 hours post dose | 0.49 [-0.23 to 1.22] | 0.73 [-0.02 to 1.48] | 0.11 [-0.82 to 1.04] | 0.58 [-0.34 to 1.51]
  Chloride, day 7, 0.0 hour | 1.46 [0.40 to 2.53] | 1.28 [0.19 to 2.37] | 0.89 [0.17 to 1.62] | 0.63 [-0.09 to 1.36]
  Chloride, day 7, 4.0 hours post dose | 0.47 [-0.96 to 1.89] | 0.22 [-1.26 to 1.69] | -0.05 [-0.86 to 0.75] | 0.28 [-0.50 to 1.07]
  Chloride, day 7, 6.0 hours post dose | 0.87 [-0.29 to 2.03] | 1.32 [0.11 to 2.52] | -0.21 [-1.00 to 0.58] | -0.86 [-1.68 to -0.04]
  Chloride, day 7, 12.0 hours post dose | 0.98 [-0.12 to 2.09] | 1.20 [0.06 to 2.35] | -1.16 [-2.08 to -0.25] | -1.48 [-2.43 to -0.53]
  Potassium, day 1, 2.0 hours post dose | 1.96 [-0.71 to 4.63] | -1.25 [-4.01 to 1.51] | -1.20 [-3.86 to 1.45] | 1.69 [-0.86 to 4.24]
  Potassium, day 1, 4.0 hours post dose | -0.16 [-3.73 to 3.41] | -0.11 [-3.80 to 3.58] | 0.42 [-6.10 to 6.95] | 1.11 [-5.17 to 7.39]
  Potassium, day 1, 6.0 hours post dose | -2.91 [-5.82 to 0.01] | -5.88 [-8.90 to -2.87] | -0.63 [-8.29 to 7.02] | -2.61 [-10.00 to 4.79]
  Potassium, day 1, 12.0 hours post dose | 6.63 [-0.02 to 13.28] | 15.27 [8.40 to 22.15] | 18.57 [10.49 to 26.64] | 19.96 [11.85 to 28.08]
  Potassium, day 2, 24.0 hours post dose | 2.06 [-1.44 to 5.56] | 0.14 [-3.48 to 3.76] | 7.70 [1.23 to 14.18] | 7.00 [0.51 to 13.49]
  Potassium, day 7, 0.0 hour | 1.06 [-2.80 to 4.93] | -1.55 [-5.55 to 2.45] | -0.47 [-4.70 to 3.76] | 1.29 [-2.93 to 5.52]
  Potassium, day 7, 4.0 hours post dose | -2.16 [-5.21 to 0.89] | -2.93 [-6.08 to 0.22] | 3.61 [-5.71 to 12.94] | 0.28 [-8.60 to 9.16]
  Potassium, day 7, 6.0 hours post dose | -3.23 [-6.47 to 0.00] | -5.16 [-8.49 to -1.84] | -4.20 [-10.85 to 2.45] | -4.14 [-11.06 to 2.78]
  Potassium, day 7, 12.0 hours post dose | 17.22 [9.58 to 24.86] | 12.32 [4.37 to 20.26] | 18.19 [7.38 to 29.01] | 19.28 [8.12 to 30.45]
  Sodium, day 1, 2.0 hours post dose | -1.09 [-1.68 to -0.50] | -0.67 [-1.28 to -0.05] | -0.63 [-1.10 to -0.16] | -0.17 [-0.63 to 0.29]
  Sodium, day 1, 4.0 hours post dose | -1.82 [-2.52 to -1.13] | -1.18 [-1.90 to -0.45] | -0.18 [-0.84 to 0.48] | -0.04 [-0.67 to 0.59]
  Sodium, day 1, 6.0 hours post dose | -1.47 [-2.09 to -0.84] | -1.12 [-1.77 to -0.47] | -0.62 [-1.20 to -0.04] | -0.17 [-0.73 to 0.39]
  Sodium, day 1, 12.0 hours post dose | -0.17 [-0.74 to 0.39] | 0.48 [-0.11 to 1.07] | -0.12 [-0.91 to 0.68] | 0.14 [-0.66 to 0.93]
  Sodium, day 2, 24.0 hours post dose | 0.03 [-0.78 to 0.84] | 1.06 [0.22 to 1.90] | 0.85 [0.24 to 1.45] | 1.24 [0.63 to 1.84]
  Sodium, day 7, 0.0 hour | 1.21 [0.23 to 2.18] | 1.36 [0.35 to 2.37] | 0.69 [0.05 to 1.33] | 0.84 [0.20 to 1.48]
  Sodium, day 7, 4.0 hours post dose | -0.25 [-1.46 to 0.95] | -0.89 [-2.14 to 0.37] | -0.81 [-1.57 to -0.05] | -0.16 [-0.89 to 0.57]
  Sodium, day 7, 6.0 hours post dose | 0.01 [-1.17 to 1.19] | -0.19 [-1.42 to 1.05] | -0.74 [-1.36 to -0.13] | -0.86 [-1.49 to -0.23]
  Sodium, day 7, 12.0 hours post dose | 0.34 [-0.62 to 1.29] | 0.78 [-0.22 to 1.77] | -0.41 [-1.23 to 0.42] | -1.04 [-1.89 to -0.20]

14. Secondary Outcome: Percent Change From Baseline in Blood Plasma Creatinine
Description: Blood plasma creatinine was analyzed at a central laboratory.
Time Frame: 4, 6 and 12 hours post dose on day 1; 24 hours post dose on day 2; 0, 4, 6 and 12 hours post dose on day 7
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | LCZ696 - Heart Failure (HF) Cohort | Valsartan - HF Cohort | LCZ696 - Hypertension (HTN) Cohort | Valsartan - HTN Cohort
Number analyzed (Participants) | 16 | 16 | 16 | 16
Percentage change
  Day 1, 4.0 hours post dose | -7.06 [-9.03 to -5.10] | -3.55 [-5.56 to -1.54] | -7.48 [-9.28 to -5.68] | -0.91 [-2.65 to 0.83]
  Day 1, 6.0 hrs post dose | -2.97 [-5.49 to -0.46] | -0.07 [-2.67 to 2.54] | -1.72 [-5.41 to 1.96] | 4.40 [0.84 to 7.95]
  Day 1, 12.0 hrs post dose | 3.02 [-1.96 to 8.00] | 5.36 [0.21 to 10.52] | 6.22 [1.90 to 10.54] | 9.23 [5.07 to 13.40]
  Day 2, 24 hrs post dose | 3.73 [-1.37 to 8.83] | 4.02 [-1.26 to 9.30] | 13.64 [8.44 to 18.84] | 6.18 [1.15 to 11.21]
  Day 7, 0.0 hour | 4.24 [-6.71 to 15.19] | 0.55 [-10.43 to 11.52] | 1.76 [-1.74 to 5.27] | 1.71 [-1.79 to 5.21]
  Day 7, 4.0 hrs post dose | -1.47 [-8.56 to 5.63] | -5.09 [-12.26 to 2.07] | -3.02 [-6.71 to 0.68] | -1.28 [-4.98 to 2.41]
  Day 7, 6.0 hrs post dose | 1.72 [-6.15 to 9.59] | -0.25 [-8.18 to 7.68] | 0.48 [-3.44 to 4.40] | 3.03 [-0.89 to 6.94]
  Day 7, 12 hrs post dose | 8.03 [-3.02 to 19.07] | 8.34 [-2.79 to 19.48] | 9.33 [4.43 to 14.24] | 4.55 [-0.35 to 9.46]

15. Secondary Outcome: Glomerular Filtration Rate (GFR) Over Time
Description: GFR was used as a measure of renal function.
Time Frame: 0, 2, 4 and 6 hours post dose on day 1; 0, 2, 4 and 6 hours post dose on day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | LCZ696 - Heart Failure (HF) Cohort | Valsartan - HF Cohort | LCZ696 - Hypertension (HTN) Cohort | Valsartan - HTN Cohort
Number analyzed (Participants) | 16 | 16 | 16 | 16
mL/min
  Day 1, 0 hour | 76.4 (43.27) | 92.5 (97.37) | 87.6 (64.27) | 99.2 (66.36)
  Day 1, 2 hours post dose | 115.7 (57.89) | 83.3 (46.57) | 112.1 (63.30) | 96.0 (44.23)
  Day 1, 4 hours post dose | 117.4 (75.09) | 70.9 (36.64) | 125.4 (95.33) | 101.8 (65.34)
  Day 1, 6 hours post dose | 120.2 (68.73) | 71.7 (37.27) | 148.4 (138.66) | 123.0 (60.62)
  Day 7, 0 hour | 93.7 (75.98) | 87.8 (57.47) | 96.8 (78.65) | 83.2 (53.11)
  Day 7, 2 hours post dose | 95.9 (39.47) | 83.1 (35.65) | 133.5 (67.82) | 91.4 (50.57)
  Day 7, 4 hours post dose | 89.6 (52.23) | 94.6 (53.43) | 151.7 (109.91) | 111.3 (59.41)
  Day 7, 6 hours post dose | 86.9 (49.26) | 126.6 (79.95) | 111.5 (66.30) | 165.2 (228.97)

16. Secondary Outcome: Renal Blood Flow (RBF) Over Time
Description: RBF was used as a measure of renal function.
Time Frame: 0, 2, 4 and 6 hours post dose on day 1; 0, 2, 4 and 6 hours post dose on day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | LCZ696 - Heart Failure (HF) Cohort | Valsartan - HF Cohort | LCZ696 - Hypertension (HTN) Cohort | Valsartan - HTN Cohort
Number analyzed (Participants) | 16 | 16 | 16 | 16
mL/min
  Day 1, 0 hour | 398.1 (221.24) | 305.7 (159.44) | 774.7 (893.23) | 737.0 (323.14)
  Day 1, 2 hours post dose | 361.3 (171.80) | 357.4 (218.28) | 570.5 (212.67) | 541.7 (179.20)
  Day 1, 4 hours post dose | 340.1 (169.87) | 297.4 (219.83) | 700.0 (408.73) | 573.4 (287.14)
  Day 1, 6 hours post dose | 465.2 (276.84) | 290.05 (138.30) | 1165.2 (912.25) | 758.7 (375.11)
  Day 7, 0 hour | 354.9 (223.49) | 417.0 (254.35) | 548.5 (389.77) | 549.3 (247.41)
  Day 7, 2 hours | 331.9 (180.59) | 341.1 (156.86) | 630.4 (239.55) | 659.1 (426.18)
  Day 7, 4 hours | 324.2 (168.10) | 285.9 (150.82) | 653.2 (412.91) | 606.3 (224.57)
  Day 7, 6 hours | 331.0 (228.38) | 440.8 (310.64) | 667.6 (308.52) | 977.9 (975.25)

17. Secondary Outcome: Supine Systolic Blood Pressure
Description: Systolic blood pressure measurements were taken.
Time Frame: 0, 0.5, 1, 2, 4, 8 and 12 hours post dose on day 1; day 2; 0, 0.5, 1, 2, 4, 8 and 12 hours post dose on day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LCZ696 - Heart Failure (HF) Cohort | Valsartan - HF Cohort | LCZ696 - Hypertension (HTN) Cohort | Valsartan - HTN Cohort
Number analyzed (Participants) | 16 | 16 | 16 | 16
mmHg
  Day 1, 0.0 hour | 114.8 (14.10) | 127.0 (16.62) | 136.1 (18.80) | 133.2 (14.79)
  Day 1, 0.5 hour post dose | 122.8 (14.36) | 121.5 (21.78) | 132.9 (19.52) | 132.5 (17.85)
  Day 1, 1.0 hour post dose | 123.9 (16.53) | 122.2 (19.20) | 134.1 (18.57) | 133.2 (15.22)
  Day 1, 2.0 hours post dose | 125.4 (13.68) | 127.2 (16.71) | 134.2 (19.85) | 132.6 (17.47)
  Day 1, 4.0 hours post dose | 133.1 (18.65) | 130.3 (17.14) | 140.7 (20.67) | 142.1 (17.93)
  Day 1, 8.0 hours post dose | 113.6 (13.29) | 120.9 (16.85) | 127.3 (17.39) | 132.2 (11.40)
  Day 1, 12.0 hours post dose | 111.1 (14.75) | 114.8 (17.85) | 127.4 (13.92) | 134.1 (14.64)
  Day 2 | 115.8 (9.61) | 120.9 (18.05) | 125.4 (12.66) | 128.9 (13.99)
  Day 7, 0.0 hour | 110.5 (10.03) | 115.9 (15.47) | 128.9 (14.83) | 128.8 (13.76)
  Day 7, 0.5 hour post dose | 116.2 (10.93) | 122.9 (11.78) | 127.4 (16.26) | 130.9 (15.06)
  Day 7, 1.0 hour post dose | 117.9 (10.01) | 124.8 (12.43) | 127.4 (17.46) | 130.9 (15.47)
  Day 7, 2.0 hours post dose | 119.3 (12.70) | 127.5 (11.95) | 128.6 (19.35) | 140.7 (15.89)
  Day 7, 4.0 hours post dose | 120.6 (11.71) | 128.9 (13.13) | 130.5 (18.15) | 134.9 (13.20)
  Day 7, 8.0 hours post dose | 111.3 (12.52) | 119.3 (10.44) | 123.1 (12.72) | 130.0 (15.88)
  Day 7, 12.0 hours post dose | 107.9 (16.70) | 116.5 (14.85) | 120.3 (12.60) | 131.9 (18.71)

18. Secondary Outcome: Supine Diastolic Blood Pressure
Description: Diastolic blood pressure measurements were taken.
Time Frame: 0, 0.5, 1, 2, 4, 8 and 12 hours post dose on day 1; day 2; 0, 0.5, 1, 2, 4, 8 and 12 hours post dose on day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LCZ696 - Heart Failure (HF) Cohort | Valsartan - HF Cohort | LCZ696 - Hypertension (HTN) Cohort | Valsartan - HTN Cohort
Number analyzed (Participants) | 16 | 16 | 16 | 16
mmHg
  Day 1, 0.0 hour | 68.2 (9.85) | 74.1 (13.20) | 77.6 (10.57) | 74.9 (9.99)
  Day 1, 0.5 hour post dose | 71.2 (12.00) | 75.5 (13.77) | 76.3 (11.85) | 75.8 (10.67)
  Day 1, 1.0 hour post dose | 71.3 (12.00) | 75.8 (13.73) | 75.3 (10.37) | 76.2 (9.59)
  Day 1, 2.0 hours post dose | 73.3 (12.01) | 77.1 (10.61) | 77.6 (11.79) | 76.0 (10.78)
  Day 1, 4.0 hours post dose | 75.6 (13.77) | 79.1 (12.21) | 80.0 (13.60) | 79.9 (9.08)
  Day 1, 8.0 hours post dose | 68.5 (11.15) | 70.4 (11.12) | 75.2 (10.23) | 76.2 (8.89)
  Day 1, 12.0 hours post dose | 65.4 (11.49) | 71.7 (13.43) | 75.5 (8.33) | 75.7 (8.81)
  Day 2 | 71.6 (10.03) | 74.9 (13.33) | 73.2 (10.78) | 75.1 (8.35)
  Day 7, 0.0 hour | 66.9 (11.04) | 68.4 (11.37) | 74.7 (8.77) | 74.7 (9.62)
  Day 7, 0.5 hour post dose | 69.6 (11.74) | 73.9 (9.48) | 74.3 (9.36) | 74.5 (9.65)
  Day 7, 1.0 hour post dose | 69.3 (10.49) | 73.9 (8.94) | 73.5 (8.52) | 75.1 (8.71)
  Day 7, 2.0 hours post dose | 70.6 (11.85) | 76.7 (9.15) | 72.0 (8.20) | 78.8 (9.29)
  Day 7, 4.0 hours post dose | 69.6 (11.17) | 74.5 (10.86) | 74.4 (9.60) | 78.4 (9.77)
  Day 7, 8.0 hours post dose | 69.3 (10.08) | 71.5 (8.43) | 71.4 (7.84) | 75.3 (8.50)
  Day 7, 12.0 hours post dose | 65.3 (10.95) | 69.8 (12.39) | 70.7 (8.36) | 75.7 (11.47)

19. Secondary Outcome: Supine Pulse Rate
Description: Pulse rate measurements were taken.
Time Frame: 0, 0.5, 1, 2, 4, 8 and 12 hours post dose on day 1; day 2; 0, 0.5, 1, 2, 4, 8 and 12 hours post dose on day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: BPM
Arm/Group | LCZ696 - Heart Failure (HF) Cohort | Valsartan - HF Cohort | LCZ696 - Hypertension (HTN) Cohort | Valsartan - HTN Cohort
Number analyzed (Participants) | 16 | 16 | 16 | 16
BPM
  Day 1, 0.0 hour | 56.8 (8.89) | 61.7 (14.30) | 65.7 (9.26) | 65.5 (8.44)
  Day 1, 0.5 hour post dose | 61.3 (9.34) | 60.7 (10.45) | 64.1 (8.59) | 63.4 (9.29)
  Day 1, 1.0 hour post dose | 62.4 (8.97) | 62.7 (10.19) | 64.2 (7.49) | 64.0 (10.39)
  Day 1, 2.0 hours post dose | 61.0 (9.02) | 64.3 (12.39) | 65.6 (8.28) | 63.2 (8.89)
  Day 1, 4.0 hours post dose | 60.0 (8.51) | 62.9 (13.29) | 64.0 (6.51) | 65.3 (9.65)
  Day 1, 8.0 hours post dose | 67.6 (11.70) | 69.1 (11.34) | 73.9 (10.20) | 67.5 (10.09)
  Day 1, 12.0 hours post dose | 61.1 (13.36) | 62.8 (10.83) | 73.7 (13.52) | 65.4 (9.68)
  Day 2 | 60.1 (12.18) | 64.5 (11.95) | 71.3 (10.58) | 66.5 (9.20)
  Day 7, 0.0 hour post dose | 63.0 (11.97) | 60.6 (12.69) | 62.9 (5.54) | 62.8 (8.16)
  Day 7, 0.5 hour post dose | 65.0 (12.63) | 60.1 (12.07) | 63.0 (4.36) | 61.8 (9.35)
  Day 7, 1.0 hour post dose | 63.3 (13.21) | 61.6 (11.70) | 62.3 (5.87) | 61.6 (7.70)
  Day 7, 2.0 hours post dose | 63.9 (10.42) | 58.7 (11.49) | 61.2 (6.17) | 63.6 (9.16)
  Day 7, 4.0 hours post dose | 65.7 (10.85) | 60.7 (11.34) | 62.9 (6.45) | 62.7 (9.20)
  Day 7, 8.0 hours post dose | 67.1 (10.20) | 66.5 (11.80) | 66.3 (7.34) | 64.8 (10.83)
  Day 7, 12.0 hours post dose | 66.7 (13.28) | 71.9 (17.30) | 66.2 (6.97) | 67.1 (11.10)

ADVERSE EVENTS:
Arm/Group | LCZ696 - Heart Failure (HF) Cohort | Valsartan - HF Cohort | LCZ696 - Hypertension (HTN) Cohort | Valsartan - HTN Cohort
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 3/16 | 1/15 | 1/15 | 3/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 - Heart Failure (HF) Cohort (N=16) | Valsartan - HF Cohort (N=15) | LCZ696 - Hypertension (HTN) Cohort (N=15) | Valsartan - HTN Cohort (N=16)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Regarding LSM = 1218.56 for LCZ696 HTN cohort arm at Day 1, 1.0 hr post dose, the value was heavily inflated due to one participant with a very high change from baseline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.